CLINICAL TRIAL: NCT01862705
Title: Using fMRI to Determine if Cerebral Hemodynamic Responses to Pain Change Following Thoracic Spine Manipulation in Individuals With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OSF Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 449272-1
Record Dates: First submitted 2013-05-09; First posted 2013-05-24 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic spine manipulation thrust (Experimental): Thoracic spine manipulation thrust
  Interventions: Other: Thoracic spine manipulation
- Thoracic spine manipulation non-thrust (Sham Comparator): Thoracic spine manipulation non-thrust
  Interventions: Other: Thoracic spine manipulation

INTERVENTIONS:
Other: Thoracic spine manipulation — TSM thrust or non-thrust

SUMMARY:
Thoracic spine thrust manipulation (TSM) has been shown to be an effective intervention in the management of patients with neck pain. However the mechanisms for pain relief associated with this intervention remain largely unexplained. Recent evidence suggests structures within the brain may have a role in creating responses of pain relief. This study aims to use functional magnetic resonance imaging (fMRI) to determine if there is a change in blood flow to structures within the brain following TSM in patients with neck pain. All patients will undergo fMRI while receiving painful stimuli directed to two separate sites, the cuticle of the index finger and the great toe. Subjects will then receive either TSM or sham-manipulation and then immediately undergo a second fMRI scan receiving the same painful stimuli. The primary outcome of interest is the shift in blood flow within the brain before and after TSM or sham manipulation as measured by Blood Oxygen Level Dependent (BOLD) technology. This study will be the first to examine this type of response to manual therapy within the brain in patients with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of mechanical neck pain of less than 6 weeks in duration as identified in the patient's initial physical examination. Mechanical neck pain is defined as generalized neck and/or shoulder, peri-scapular pain with symptoms provoked by neck postures, neck movements, or palpation of the cervical musculature

Exclusion Criteria:

* Any medical red flags suggestive of non-musculoskeletal origin of pain, such as metabolic disorders, osteoporosis, tumor, and/or rheumatoid arthritis
* No contraindications to spinal mobilization
* No contraindications to MRI (claustrophobia, presence of cardiac pacemakers, cochlear implants, metal implants, implanted hearing aids, and previous injuries caused by bullets or shrapnel, pregnancy or thought to be pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
BOLD response to noxious stimuli | Immediately following TSM or sham-manipulation. Time frame to initiate MR scanning following thrust or sham-manipulation not to exceed 5 minutes.
  shift in blood flow within the brain before and after TSM or sham manipulation as measured by Blood Oxygen Level Dependent (BOLD) technology, as measured by fMRI.

CONTACTS AND LOCATIONS:
Locations (1):
- OSF Saint Francis Medical Center, Peoria, Illinois, United States